CLINICAL TRIAL: NCT04520659
Title: Phase Ib Placebo-Controlled Study of the Infectivity, Safety and Immunogenicity of a Single Dose of a Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine, LID/ΔM2-2/1030s, Lot RSV#010A, Delivered as Nose Drops to RSV-Seronegative Infants and Children 6 to 24 Months of Age
Brief Title: Evaluating the Infectivity, Safety and Immunogenicity of a Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine, LID/ΔM2-2/1030s, in RSV-Seronegative Infants and Children 6 to 24 Months of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 335
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: RSV LID/ΔM2-2/1030s (Experimental): Participants will receive a single dose of RSV LID/ΔM2-2/1030s vaccine at study entry (Day 0).
  Interventions: Biological: RSV LID/ΔM2-2/1030s
- Group 1: Placebo (Placebo Comparator): Participants will receive a single dose of placebo at study entry (Day 0).
  Interventions: Biological: Placebo
- Group 2: RSV LID/ΔM2-2/1030s (Experimental): Participants will receive a single dose of RSV LID/ΔM2-2/1030s vaccine at study entry (Day 0).
  Interventions: Biological: RSV LID/ΔM2-2/1030s
- Group 2: Placebo (Placebo Comparator): Participants will receive a single dose of placebo at study entry (Day 0).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV LID/ΔM2-2/1030s — 10^5 plaque-forming units (PFU); administered as nose drops
  Arms: Group 1: RSV LID/ΔM2-2/1030s; Group 2: RSV LID/ΔM2-2/1030s
Biological: Placebo — Administered as nose drops
  Arms: Group 1: Placebo; Group 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the infectivity, safety, and immunogenicity of a single dose of a recombinant, live-attenuated respiratory syncytial virus (RSV) vaccine, LID/ΔM2-2/1030s, in RSV-seronegative infants and children 6 to 24 months of age.

DETAILED DESCRIPTION:
This study will evaluate the infectivity, safety, and immunogenicity of a single dose of a recombinant, live-attenuated respiratory syncytial virus (RSV) vaccine, LID/ΔM2-2/1030s, in RSV-seronegative infants and children 6 to 24 months of age.

Participants will be randomly assigned to one of two groups to receive a single dose of intranasal RSV LID/ΔM2-2/1030s vaccine or placebo at study entry (Day 0). Group 1 (intensive) and Group 2 (less intensive) will differ only in the frequency of study visits and nasal swab collections.

Participants will receive study product between April 1 and October 15, outside of the RSV season, and will remain on the study until they complete the post-RSV season visit between April 1 and April 30 in the calendar year following enrollment. Participants' total study duration is between 6 and 13 months, depending upon time of enrollment.

Participants will attend several study visits throughout the study, which may include blood collection, nasal swabs, and physical examinations. Some of these visits may be remote if a stay at home order is put in place after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 months of age and <25 months of age at the time of inoculation
* Screening and pre-inoculation serum specimens for respiratory syncytial virus (RSV)-neutralizing antibody are obtained no more than 42 days prior to inoculation
* Seronegative for RSV antibody, defined as serum RSV-neutralizing antibody titer <1:40
* In good health based on review of the medical record, history, and physical examination at the time of inoculation
* Received routine immunizations appropriate for age based on the Advisory Committee on Immunization Practices (ACIP) Recommended Immunization Schedule for Children and Adolescents Aged 18 Years or Younger
* Growing normally for age as demonstrated on a World Health Organization (WHO) growth chart, AND

  * If < 1 year of age: has a current height and weight above the 5th percentile for age
  * If ≥ 1 year of age: has a current height and weight above the 3rd percentile for age
* Expected to be available for the duration of the study
* Parent/guardian is willing and able to provide written informed consent

Exclusion Criteria:

* ≤ 6 months of age and > 25 months of age at the time of inoculation
* Born at less than 34 weeks gestation
* Born at less than 37 weeks gestation, and at the date of inoculation less than 1 year of age
* Maternal history of a positive HIV test before or during pregnancy
* Evidence of chronic disease
* Known or suspected infection or impairment of immunological functions
* Bone marrow/solid organ transplant recipient
* Major congenital malformations, including congenital cleft palate or cytogenetic abnormalities
* Suspected or documented developmental disorder, delay, or other developmental problem
* Cardiac abnormality requiring treatment
* Lung disease or reactive airway disease
* More than one episode of medically diagnosed wheezing in the first year of life
* Wheezing episode or received bronchodilator therapy within the past 12 months
* Wheezing episode or received bronchodilator therapy after the age of 12 months
* Previous receipt of supplemental oxygen therapy in a home setting
* Previous receipt of an investigational RSV vaccine
* Previous receipt or planned administration of anti-RSV antibody product including ribavirin, RSV Ig, or RSV mAb
* Previous receipt of immunoglobulin or any antibody products within the past 6 months
* Previous receipt of any blood products within the past 6 months
* Previous anaphylactic reaction
* Previous vaccine-associated adverse reaction that was Grade 3 or above
* Known hypersensitivity to any study product component
* Member of a household that contains an infant who is less than 6 months of age at the date of inoculation through the 28th day after inoculation
* Member of a household that, at the date of inoculation through the 28th day after inoculation, contains an immunocompromised individual including but not limited to:

  * a person who is HIV-infected
  * a person who has cancer and has received chemotherapy within the 12 months prior to enrollment
  * a person living with a solid organ or bone marrow transplant
* Attends a daycare facility that does not separate children by age and contains an infant <6 months of age at the date of inoculation through the 28th day after inoculation
* Receipt of any of the following prior to enrollment:

  * inactivated influenza vaccine within 3 days prior, or
  * any other inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior, or
  * salicylate (aspirin) or salicylate-containing products within the past 28 days
* Scheduled administration of any of the following after planned inoculation

  * inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days after, or
  * any live vaccine other than rotavirus in the 28 days after, or
  * another investigational vaccine or investigational drug in the 56 days after
* Receipt of any of the following medications within 3 days of study enrollment:

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medications except the permitted concomitant medications listed below
* Permitted concomitant medications (prescription or non-prescription) include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) cutaneous (topical) steroids, topical antibiotics, and topical antifungal agents.
* Any of the following events at the time of enrollment:

  * fever (temporal or rectal temperature of ≥100.4°F), or
  * upper respiratory signs or symptoms (rhinorrhea, cough, or pharyngitis) or
  * nasal congestion significant enough to interfere with successful inoculation, or
  * otitis media
  * contact with a person diagnosed with COVID-19 disease or active severe acute respiratory syndrome coronavirus 2 (SARS CoV-2) infection within the preceding 10 days

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health (JHSPH)
Locations (3):
- United States (3):
  - John Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - University of Rochester Medical Center, Rochester, New York
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to IPD that underlie results in a publication. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants.
Time Frame: After publication
Access Criteria: Qualified researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from pediatric practices and clinics in the greater Baltimore, MD/Washington, DC, Rochester, NY and Nashville, TN areas based on referral by the primary care provider or the provider's staff; and through electronic patient portals using IRB-approved messages. These recruitment methods targeted age-appropriate children between February, 2022 and March, 2023. The first participant was enrolled on 3/16/22 and the last participant was enrolled on 5/10/23.
Pre-assignment Details: Of the 111 participants that were screened, 81 met eligibility criteria and the parent agreed to enroll their child. The 81 children were then inoculated with study product.
Period: Acute Phase (Days 0-28)
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 1: Placebo | Group 2: RSV LID/ΔM2-2/1030s | Group 2: Placebo
Started | 14 | 7 | 40 | 20
Completed | 14 | 7 | 40 | 20
Not Completed | 0 | 0 | 0 | 0
Period: RSV Surveillance Phase Oct. 16-March 31
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 1: Placebo | Group 2: RSV LID/ΔM2-2/1030s | Group 2: Placebo
Started | 14 | 7 | 40 | 20
Completed | 13 | 7 | 39 | 20
Not Completed | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 1: Placebo | Group 2: RSV LID/ΔM2-2/1030s | Group 2: Placebo | Total
Number analyzed (Participants) | 14 | 7 | 40 | 20 | 81
Age, Customized [Count of Participants; unit: Participants]
  < 6 months of age | 0 | 0 | 0 | 0 | 0
  6-12 months of age | 8 | 1 | 25 | 8 | 42
  13-18 months of age | 3 | 2 | 10 | 9 | 24
  19-24 months of age | 3 | 4 | 5 | 3 | 15
  > 24 months of age | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 19 | 9 | 41
  Male | 4 | 4 | 21 | 11 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 6 | 2 | 10
  Not Hispanic or Latino | 12 | 7 | 33 | 18 | 70
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 11 | 7 | 37 | 18 | 73
  More than one race | 1 | 0 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 7 | 40 | 20 | 81

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Grade 1 or Higher Solicited Adverse Events (AEs) by Grade
Description: Solicited adverse events include fever; otitis media; upper respiratory illness (URI); lower respiratory illness (LRI) and cough (without LRI) as defined in Appendix III of the protocol document. The number of participants who experienced solicited adverse events was presented. A participant was only counted once in each solicited AE category, and that is in the line corresponding to the highest grade adverse event they had in that category. These events were graded (Grade 1-mild to Grade 4-life-threatening) following protocol-defined grading system outlined in Table 16 and Table 17 in the protocol document. Details regarding LRIs will be noted in Primary Outcome Measure #2.
Time Frame: Measured through Day 28
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Groups:
- Groups 1 and 2 Combined: RSV LID/ΔM2-2/1030s: Participants will receive a single dose of RSV LID/ΔM2-2/1030s vaccine at study entry (Day 0).
  RSV LID/ΔM2-2/1030s: 10^5 plaque-forming units (PFU); administered as nose drops
- Groups 1 and 2 Combined: Placebo: Participants will receive a single dose of placebo at study entry (Day 0).
  Placebo: Administered as nose drops
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 1: Placebo | Group 2: RSV LID/ΔM2-2/1030s | Group 2: Placebo | Groups 1 and 2 Combined: RSV LID/ΔM2-2/1030s | Groups 1 and 2 Combined: Placebo
Number analyzed (Participants) | 14 | 7 | 40 | 20 | 54 | 27
Participants
  Fever: Did not have this AE | 14 | 7 | 27 | 11 | 41 | 18
  Fever: Grade 1 | 0 | 0 | 8 | 4 | 8 | 4
  Fever: Grade 2 | 0 | 0 | 4 | 1 | 4 | 1
  Fever: Grade 3 | 0 | 0 | 1 | 3 | 1 | 3
  Fever: Grade 4 | 0 | 0 | 0 | 1 | 0 | 1
  Upper Respiratory: Did not have this AE | 4 | 4 | 13 | 12 | 17 | 16
  Upper Respiratory: Grade 1 | 9 | 3 | 24 | 7 | 33 | 10
  Upper Respiratory: Grade 2 | 1 | 0 | 3 | 1 | 4 | 1
  Upper Respiratory: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Upper Respiratory: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Did not have this AE | 14 | 7 | 39 | 20 | 53 | 27
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 2 | 0 | 0 | 1 | 0 | 1 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  LRI in the absence of RSV shedding: Did not have this AE | 14 | 7 | 40 | 20 | 54 | 27
  LRI in the absence of RSV shedding: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  LRI in the absence of RSV shedding: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  LRI in the absence of RSV shedding: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  LRI in the absence of RSV shedding: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Cough without LRI: Did not have this AE | 11 | 6 | 29 | 16 | 40 | 22
  Cough without LRI: Grade 1 | 2 | 0 | 9 | 3 | 11 | 3
  Cough without LRI: Grade 2 | 1 | 1 | 2 | 1 | 3 | 2
  Cough without LRI: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Cough without LRI: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Otitis media: Did not have this AE | 14 | 7 | 37 | 18 | 51 | 25
  Otitis media: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Otitis media: Grade 2 | 0 | 0 | 3 | 2 | 3 | 2
  Otitis media: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Otitis media: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Frequency of Grade 2 or Higher Lower Respiratory Infections (LRI) by Grade
Description: LRI may include wheezing, pneumonia, laryngotracheobronchitis (croup), rhonchi and rales as defined in Appendix III of the protocol document. A participant was only counted once in each LRI category, and that is in the line corresponding to the highest grade adverse event they had in that category. These events were graded (Grade 1-mild to Grade 4-life-threatening) following protocol-defined grading system outlined in Table 16 and Table 17 in the protocol document.
Time Frame: Measured through Day 28
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 1: Placebo | Group 2: RSV LID/ΔM2-2/1030s | Group 2: Placebo | Groups 1 and 2 Combined: RSV LID/ΔM2-2/1030s | Groups 1 and 2 Combined: Placebo
Number analyzed (Participants) | 14 | 7 | 40 | 20 | 54 | 27
Participants
  Wheezing: Did not have this LRI | 14 | 7 | 40 | 20 | 54 | 27
  Wheezing: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Wheezing: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Wheezing: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Wheezing: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Pneumonia: Did not have this LRI | 14 | 7 | 40 | 20 | 54 | 27
  Pneumonia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Pneumonia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Pneumonia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Pneumonia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Laryngotracheobronchitis (Croup): Did not have this LRI | 14 | 7 | 39 | 20 | 53 | 27
  Laryngotracheobronchitis (Croup): Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Laryngotracheobronchitis (Croup): Grade 2 | 0 | 0 | 1 | 0 | 1 | 0
  Laryngotracheobronchitis (Croup): Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Laryngotracheobronchitis (Croup): Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Rhonchi: Did not have this LRI | 14 | 7 | 40 | 20 | 54 | 27
  Rhonchi: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Rhonchi: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Rhonchi: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Rhonchi: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Rales: Did not have this LRI | 14 | 7 | 40 | 20 | 54 | 27
  Rales: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Rales: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Rales: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Rales: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs) by Grade of Severity
Description: Unsolicited adverse events were other events, not included in the solicited AEs. The number of participants who experienced unsolicited adverse events was presented.
Time Frame: Measured through Day 28
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 1: Placebo | Group 2: RSV LID/ΔM2-2/1030s | Group 2: Placebo | Groups 1 and 2 Combined: RSV LID/ΔM2-2/1030s | Groups 1 and 2 Combined: Placebo
Number analyzed (Participants) | 14 | 7 | 40 | 20 | 54 | 27
Participants
  Nasal Congestion: Did not have this | 14 | 6 | 29 | 18 | 43 | 24
  Nasal Congestion: Grade 1 | 0 | 1 | 11 | 2 | 11 | 3
  Nasal Congestion: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Nasal Congestion: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Nasal Congestion: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Emesis: Did not have this | 12 | 7 | 37 | 20 | 49 | 27
  Emesis: Grade 1 | 1 | 0 | 3 | 0 | 4 | 0
  Emesis: Grade 2 | 1 | 0 | 0 | 0 | 1 | 0
  Emesis: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Emesis: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea: Did not have this | 13 | 6 | 37 | 19 | 50 | 25
  Diarrhea: Grade 1 | 0 | 1 | 3 | 1 | 3 | 2
  Diarrhea: Grade 2 | 1 | 0 | 0 | 0 | 1 | 0
  Diarrhea: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Conjunctivitis: Did not have this | 12 | 7 | 40 | 19 | 52 | 26
  Conjunctivitis: Grade 1 | 1 | 0 | 0 | 0 | 1 | 0
  Conjunctivitis: Grade 2 | 1 | 0 | 0 | 1 | 1 | 1
  Conjunctivitis: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Conjunctivitis: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Pain: Did not have this | 14 | 6 | 40 | 19 | 54 | 25
  Pain: Grade 1 | 0 | 1 | 0 | 1 | 0 | 2
  Pain: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Pain: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Pain: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Did not have this | 13 | 7 | 39 | 19 | 52 | 26
  Rash: Grade 1 | 1 | 0 | 1 | 1 | 2 | 1
  Rash: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Rash: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Urinary tract infection: Did not have this | 14 | 7 | 39 | 20 | 53 | 27
  Urinary tract infection: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urinary tract infection: Grade 2 | 0 | 0 | 1 | 0 | 1 | 0
  Urinary tract infection: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Urinary tract infection: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Who Experienced Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is an AE, whether considered related to the study product or not, that:
  Results in death during the period of protocol-defined surveillance; Is life threatening: defined as an event in which the patient was at immediate risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death were it more severe; Requires inpatient hospitalization (or prolongation of existing hospitalization): defined as at least an overnight stay in the hospital or emergency ward for treatment that would have been inappropriate if administered in the outpatient setting; Results in a persistent or significant disability/incapacity; Is a congenital anomaly or birth defect, OR Is an important medical event that may not be immediately life threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
Time Frame: Measured Day 0 through Day 56 after inoculation and During the RSV Surveillance Season (Date of seasonal pause in enrollment in year of inoculation through March 31)
Population: Study participants who received inoculation and were followed on study past Day 0 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 1: Placebo | Group 2: RSV LID/ΔM2-2/1030s | Group 2: Placebo | Groups 1 and 2 Combined: RSV LID/ΔM2-2/1030s | Groups 1 and 2 Combined: Placebo
Number analyzed (Participants) | 14 | 7 | 40 | 20 | 54 | 27
Participants | 1 | 0 | 0 | 0 | 1 | 0

5. Primary Outcome: Percentage of Vaccinees With a ≥4-fold Rise in Serum RSV-neutralizing Antibody Titer
Description: Serum RSV-neutralizing antibody titers were assessed by 60% RSV-plaque reduction neutralization titer (RSV-PRNT) assay. Antibody responses were defined as a greater than or equal to 4-fold increase in titer in paired specimens, between pre-inoculation and post-inoculation time points.
Time Frame: Measured at Day 0 and Day 56
Population: Study participants who received RSV LID/ΔM2-2/1030s at inoculation and were followed on study past Day 56 were included. One study participant in Group 2 withdrew prior to the Day 56 serum collection and is not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 2: RSV LID/ΔM2-2/1030s | Groups 1 and 2 Combined: RSV LID/ΔM2-2/1030s
Number analyzed (Participants) | 14 | 39 | 53
Participants | 12 | 26 | 38

6. Primary Outcome: Peak Titer of Vaccine Virus Shed by Reverse Transcription Polymerase Chain Reaction (RT-qPCR) (Group 1 Only)
Description: This is the mean of the highest value per participant of the titer of vaccine virus shed. It was measured by RT-qPCR. Group 1 participants only. Only participants who met the definition of infection with vaccine virus were included.
Time Frame: Measured at Days 5, 7, 10, 12 and additional illness visits between Days 0 and 28.
Population: Only participants who met the definition of infection with vaccine virus were included.
Measure: Mean (Standard Deviation); unit: log 10 copies/mL
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 1: Placebo
Number analyzed (Participants) | 14 | 0
log 10 copies/mL | 6.6 (1.3) |

7. Primary Outcome: Number of Vaccinees Infected With RSV Vaccine Virus in Group 1
Description: Defined as shedding vaccine virus, detected by RT-qPCR, and/or ≥4-fold rise in RSV-specific serum antibodies, detected by enzyme-linked immunosorbent assay (ELISA) against the RSV F protein and/or an RSV-PRNT from study entry to Study Day 56
Time Frame: Measured through Day 56
Population: Study participants in Group 1 who received RSV LID/ΔM2-2/1030s at inoculation and were followed on study past Day 56 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s
Number analyzed (Participants) | 14
Participants | 14

8. Secondary Outcome: Frequency of RSV-medically Attended Acute Respiratory Illness (MAARI) by Grade in Vaccine and Placebo Recipients Who Experience Natural Infection With Wild Type RSV During the Subsequent RSV Season
Description: The number of participants who had RSV-associated, symptomatic, medically attended respiratory and febrile illness (MAARI) among those who had indicators of natural infection with wt RSV were presented. Natural infection with wt RSV during the RSV season surveillance was defined as having either RSV detected in nasal swabs collected during illness visits for MAARI events or a > 2.5-fold rise in serum antibodies from pre- to post-RSV season in the absence of RSV-associated medical events. A participant was only counted once in each solicited AE category, and that is in the line corresponding to the highest grade adverse event they had in that category. These events were graded (Grade 1-mild to Grade 4-life-threatening) following protocol-defined grading system outlined in Table 16 and Table 17 in the protocol document.
Time Frame: Measured during RSV season (from date of seasonal pause in enrollment in the year of inoculation through March 31)
Population: Only participants who had RSV detected in nasal swabs or had > 4 fold rise in serum antibodies from pre- to post-RSV season in the absence of RSV-associated medical events were included. Two vaccinees were excluded due to withdrawing prior to the completing the RSV surveillance period, and one placebo recipient was excluded due to parent refused to allow collection of the post-surveillance serum sample. Medically Attended Lower Respiratory Illness will be detailed in Secondary Outcome #9
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 1: Placebo | Group 2: RSV LID/ΔM2-2/1030s | Group 2: Placebo | Groups 1 and 2 Combined: RSV LID/ΔM2-2/1030s | Groups 1 and 2 Combined: Placebo
Number analyzed (Participants) | 13 | 5 | 27 | 11 | 40 | 16
Participants
  Fever: Did not have this MAARI | 8 | 4 | 15 | 7 | 23 | 11
  Fever: Grade 1 | 0 | 0 | 3 | 1 | 3 | 1
  Fever: Grade 2 | 0 | 0 | 3 | 2 | 3 | 2
  Fever: Grade 3 | 5 | 1 | 6 | 1 | 11 | 2
  Fever: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Upper Respiratory Illness: Did not have this MAARI | 6 | 2 | 12 | 4 | 18 | 6
  Upper Respiratory Illness: Grade 1 | 0 | 0 | 0 | 2 | 0 | 2
  Upper Respiratory Illness: Grade 2 | 7 | 3 | 15 | 5 | 22 | 8
  Upper Respiratory Illness: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Upper Respiratory Illness: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Lower Respiratory Illness with RSV: Did not have this MAARI | 11 | 5 | 26 | 10 | 37 | 15
  Lower Respiratory Illness with RSV: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Lower Respiratory Illness with RSV: Grade 2 | 1 | 0 | 1 | 1 | 2 | 1
  Lower Respiratory Illness with RSV: Grade 3 | 1 | 0 | 0 | 0 | 1 | 0
  Lower Respiratory Illness with RSV: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  LRI in the absence of RSV: Did not have this MAARI | 11 | 5 | 25 | 11 | 36 | 16
  LRI in the absence of RSV: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  LRI in the absence of RSV: Grade 2 | 2 | 0 | 2 | 0 | 4 | 0
  LRI in the absence of RSV: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  LRI in the absence of RSV: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Cough without LRI: Did not have this MAARI | 8 | 2 | 12 | 5 | 20 | 7
  Cough without LRI: Grade 1 | 0 | 1 | 0 | 1 | 0 | 2
  Cough without LRI: Grade 2 | 5 | 2 | 15 | 5 | 20 | 7
  Cough without LRI: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Cough without LRI: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Otitis media: Did not have this MAARI | 8 | 5 | 16 | 8 | 24 | 13
  Otitis media: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Otitis media: Grade 2 | 5 | 0 | 11 | 3 | 16 | 3
  Otitis media: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Otitis media: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Frequency of RSV-medically Attended Acute Lower Respiratory Illness (MAALRI) by Grade in Vaccine and Placebo Recipients Who Experience Natural Infection With Wild Type RSV During the Subsequent RSV Season
Description: The number of participants who had RSV-associated, symptomatic, medically attended acute lower respiratory illness (MAALRI) among those who had indicators of natural infection with wt RSV were presented. Natural infection with wt RSV during the RSV season surveillance was defined as having either RSV detected in nasal swabs collected during illness visits for MAALRI events or a ≥ 2.5-fold rise in serum antibodies from pre- to post-RSV season in the absence of RSV-associated medical events. A participant was only counted once in each LRI category, and that is in the line corresponding to the highest grade adverse event they had in that category. These events were graded (Grade 1-mild to Grade 4-life-threatening) following protocol-defined grading system outlined in Table 16 and Table 17 in the protocol document.
Time Frame: Measured during RSV season (from date of seasonal pause in enrollment in the year of inoculation through March 31)
Population: Only participants who had RSV detected in nasal swabs or had > 4 fold rise in serum antibodies from pre- to post-RSV season in the absence of RSV-associated medical events were included. Two vaccinees were excluded due to withdrawing prior to the completing the RSV surveillance period, and one placebo recipient was excluded due to parent refused to allow collection of the post-surveillance serum sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 1: Placebo | Group 2: RSV LID/ΔM2-2/1030s | Group 2: Placebo | Groups 1 and 2 Combined: RSV LID/ΔM2-2/1030s | Groups 1 and 2 Combined: Placebo
Number analyzed (Participants) | 13 | 5 | 27 | 11 | 40 | 16
Participants
  Wheezing: Did not have this MAALRI | 12 | 5 | 26 | 11 | 38 | 16
  Wheezing: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Wheezing: Grade 2 | 0 | 0 | 1 | 0 | 1 | 0
  Wheezing: Grade 3 | 1 | 0 | 0 | 0 | 1 | 0
  Wheezing: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Pneumonia: Did not have this MAALRI | 12 | 5 | 26 | 11 | 38 | 16
  Pneumonia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Pneumonia: Grade 2 | 1 | 0 | 1 | 0 | 2 | 0
  Pneumonia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Pneumonia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Bronchitis: Did not have this MAALRI | 12 | 5 | 27 | 11 | 39 | 16
  Bronchitis: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Bronchitis: Grade 2 | 1 | 0 | 0 | 0 | 1 | 0
  Bronchitis: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Bronchitis: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  laryngotracheobronchitis (Croup): Did not have this MAALRI | 11 | 5 | 26 | 11 | 37 | 16
  laryngotracheobronchitis (Croup): Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  laryngotracheobronchitis (Croup): Grade 2 | 2 | 0 | 1 | 0 | 3 | 0
  laryngotracheobronchitis (Croup): Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  laryngotracheobronchitis (Croup): Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Rhonchi: Did not have this MAALRI | 13 | 5 | 27 | 11 | 40 | 16
  Rhonchi: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Rhonchi: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Rhonchi: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Rhonchi: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Rales: Did not have this MAALRI | 13 | 5 | 26 | 11 | 39 | 16
  Rales: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Rales: Grade 2 | 0 | 0 | 1 | 0 | 1 | 0
  Rales: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Rales: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Bronchiolitis: Did not have this MAALRI | 13 | 5 | 27 | 10 | 40 | 15
  Bronchiolitis: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  Bronchiolitis: Grade 2 | 0 | 0 | 0 | 1 | 0 | 1
  Bronchiolitis: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Bronchiolitis: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Percentage of Vaccinees With a ≥4-fold Rise in Serum RSV preF IgG and/or RSV postF IgG
Description: Serum RSV preF IgG titers and RSV postF IgG titers were assessed by an Enzyme-linked Immunosorbent Assay (ELISA). Antibody responses were defined as a ≥4-fold increase in titer in paired specimens, between pre-inoculation and post-inoculation time points.
Time Frame: Measured at Day 0 and Day 56
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 2: RSV LID/ΔM2-2/1030s | Groups 1 and 2 Combined: RSV LID/ΔM2-2/1030s
Number analyzed (Participants) | 14 | 39 | 53
Participants
  RSV PreF IgG | 9 | 22 | 31
  RSV PostF IgG | 12 | 28 | 40

ADVERSE EVENTS:
Time Frame: From study entry to end of study. The duration of follow-up for a given participant was between 6 and 13 months for both Groups 1 & 2 depending on time of enrollment.
Description: From day 0-28, all SAEs, solicited AEs, and unsolicited AEs, with the exception of the following if not treated with prescription medication or over the counter medications with antipyretic properties: diaper rashes, teething pain, and spitting up. SAEs and LRIs were reported according to Sections 7 & 8 in the Protocol Document. From day 29-56, SAEs were collected. After day 56, from November 1 - March 31 of the following year, medically attended fever, LRI, URI and otitis media were collected.
Arm/Group | Group 1: RSV LID/ΔM2-2/1030s | Group 1: Placebo | Group 2: RSV LID/ΔM2-2/1030s | Group 2: Placebo | Groups 1 and 2 Combined: RSV LID/ΔM2-2/1030s | Groups 1 and 2 Combined: Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/7 | 0/40 | 0/20 | 0/54 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/7 | 0/60 | 0/20 | 1/74 | 0/27
Other Adverse Events (participants affected / at risk) | 11/14 | 4/7 | 29/40 | 14/20 | 40/54 | 18/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: RSV LID/ΔM2-2/1030s (N=14) | Group 1: Placebo (N=7) | Group 2: RSV LID/ΔM2-2/1030s (N=60) | Group 2: Placebo (N=20) | Groups 1 and 2 Combined: RSV LID/ΔM2-2/1030s (N=74) | Groups 1 and 2 Combined: Placebo (N=27)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — During RSV Surveillance Period, wheezing started on Study Day 206. Child hospitalized for 25 hours and diagnosed with RSV. Symptom resolved on Study Day 212.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: RSV LID/ΔM2-2/1030s (N=14) | Group 1: Placebo (N=7) | Group 2: RSV LID/ΔM2-2/1030s (N=40) | Group 2: Placebo (N=20) | Groups 1 and 2 Combined: RSV LID/ΔM2-2/1030s (N=54) | Groups 1 and 2 Combined: Placebo (N=27)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0) | 3 (3) | 0 (0) | 5 (7) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 13 (16) | 9 (13) | 13 (16) | 9 (13)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 11 (14) | 4 (6) | 14 (17) | 5 (7)
Croup (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 11 (13) | 2 (4) | 11 (13) | 3 (5)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 3 (3) | 27 (36) | 8 (10) | 37 (51) | 11 (13)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT04520659/Prot_SAP_001.pdf
  • Informed Consent Form: Group 1 (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT04520659/ICF_002.pdf
  • Informed Consent Form: Group 2 (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT04520659/ICF_003.pdf